CLINICAL TRIAL: NCT06144164
Title: A Prospective Cohort Study of Patients Undergoing ALND for Treatment of Breast Cancer: The Efficacy of a Comprehensive Prevention Program in Decreasing the Incidence of Lymphedema and Improving Quality of Life
Brief Title: A Study of a Comprehensive Prevention Program to Reduce Lymphedema After Axillary Lymph Node Dissection in People With Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 23-303
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Lymphedema; Lymphedema Arm; Lymphedema of Upper Arm; Breast Cancer; Breast Carcinoma; Female Breast Cancer
Keywords: immediate lymphatic reconstruction; axillary lymph node dissection; Lymphedema; Lymphedema Arm; Lymphedema of Upper Arm; Breast cancer; breast carcinoma; female breast cancer; Memorial Sloan Kettering Cancer Center; 23-303
MeSH Terms: conditions — Lymphedema; Breast Neoplasms | interventions — Manual Lymphatic Drainage; Range of Motion, Articular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants with Breast Cancer (Experimental): Participants will have a diagnosis of breast cancer and may undergo axillary lymph node dissection.
  Interventions: Procedure: Immediate Lymphatic Reconstruction; Diagnostic Test: Volumetric arm measurements; Other: Lymphatic massage; Other: Range of motion exercises; Other: Compression garment use

INTERVENTIONS:
Procedure: Immediate Lymphatic Reconstruction — Immediate Lymphatic Reconstruction will happen at the time of Axillary Lymph Node Dissection
  Other Names: ILR
Diagnostic Test: Volumetric arm measurements — Volumetric arm measurements will occur at each in-person postoperative visit time points.
Other: Lymphatic massage — Participants will begin self-directed lymphatic massage 24 to 48 h after surgery and will continue to do lymphatic massage 3 times a week for 3 months after surgery or until 3 months after any adjuvant treatments (chemotherapy, radiation, etc.) are completed
Other: Range of motion exercises — Participants will begin self-directed lymphatic massage 24 to 48 h after surgery and will continue to do lymphatic massage 3 times a week for 3 months after surgery or until 3 months after any adjuvant treatments (chemotherapy, radiation, etc.) are completed
Other: Compression garment use — Participants will use compression garments 24 to 48 h after surgery and will continue daily use for at least 8 h a day for 3 months or until 3 months after any adjuvant treatments are completed

SUMMARY:
The purpose of this study to test whether a comprehensive program may help the lymph fluid to drain out of the arm and prevent lymphedema in participants with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Diagnosis of breast cancer
* Ages 18 to 75 years
* Consented for unilateral ALND or for unilateral SLNB with possible ALND

Exclusion Criteria:

* Male sex
* Does not speak English
* Does not fit into study garment
* Axillary recurrence
* History of ALND
* Requirement of bilateral ALND for the treatment of breast cancer
* Treatment with SLNB only
* Known anaphylactic allergy to ICG dye used in ILR
* Impaired decision-making capacity

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2030-03-16 (Estimated); Study Completion 2030-03-16 (Estimated)

PRIMARY OUTCOMES:
The difference between the baseline and postoperative arm volume measurement | Up to 24 months
  The primary objective is to determine the efficacy of a prevention program in decreasing the development of lymphedema in participants treated for breast cancer with Axillary Lymph Node Dissection/ALND by use of arm volume measurements. A ≥ 10% increase in RVC (arm volume difference between the affected and unaffected arms) between baseline and postoperative measures occurring at 12 months or later will indicate the development of lymphedema

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Coriddi, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.
URL: https://www.mskcc.org

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org